CLINICAL TRIAL: NCT00553696
Title: A Phase 1 Study Of Sunitinib In Combination With S-1 And Cisplatin In Patients With Advanced Or Metastatic Gastric Cancer
Brief Title: Study Of Sunitinib With S-1 And Cisplatin For Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181127
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Stomach Neoplasms
Keywords: chemotherapy; combination
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; S 1 (combination); Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Cisplatin; Drug: S-1; Drug: Sunitinib

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 60 mg/m2 on day 1 of each 28 day cycle
Drug: S-1 — S-1 80 mg/m2 on days 1-21 of each 28 day cycle
Drug: Sunitinib — Sunitinib 25 mg, 37.5 mg and 50 mg daily S-1 80 mg/m2 on days 1-21 of each 28 day cycle Cisplatin 60 mg/m2 on day 1 of each 28 day cycle

SUMMARY:
To assess the maximal tolerated dose (MTD) and overall safety of sunitinib when administered in combination with S-1 and Cisplatin in patients with advanced/metastatic gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of gastric cancer
* Chemonaive patients
* Adequate organ function

Exclusion Criteria:

* Patients who meet the contra-indications of S-1 and Cisplatin.
* Prior chemotherapy failure patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Japan (3):
  - Aichi cancer center central hospital / Medical Oncology, Nagoya, Aichi-ken
  - Saku Central Hospital, GI Devision, Saku, Nagano
  - Shizuoka Cancer Center, Suntougun, Shizuoka

REFERENCES:
- [Derived] Boku N, Muro K, Machida N, Hashigaki S, Kimura N, Suzuki M, Lechuga M, Miyata Y. Phase I study of sunitinib plus S-1 and cisplatin in Japanese patients with advanced or metastatic gastric cancer. Invest New Drugs. 2014 Apr;32(2):261-70. doi: 10.1007/s10637-013-9948-5. Epub 2013 May 12. PMID 23665950

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three to 6 participants at each dose regimen were to be initially assessed for dose limiting toxicity (dose escalation cohort) and 10 participants were added to the maximum tolerated dose (MTD) group after MTD was determined at Sunitinib 25 mg once daily for 2 weeks followed by 2 weeks off-treatment (Schedule 2/2) regimen (MTD expansion cohort).
Groups:
- Sunitinib 25 mg CDD + S-1 + Cisplatin: Study drugs were administered at following regimens in repeating 4 week cycles; Sunitinib at dose of 25 mg orally once daily continuously (CDD), S-1 at the starting dose of 80-120 mg/day based on body surface area as a twice daily for 3 weeks followed by 1 week off-treatment, cisplatin was administered once at 60 mg/m^2 on Day 1 of each 4 week cycle.
- Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All): Study drugs were administered at following regimens in repeating 4 week cycles; Sunitinib at dose of 25 mg orally once daily for 2 weeks followed by 2 weeks off-treatment (Schedule 2/2), S-1 at the starting dose of 80-120 mg/day based on body surface area as a twice daily for 3 weeks followed by 1 week off-treatment, cisplatin was administered once at 60 mg/m^2 on Day 1 (dose escalation cohort) or Day 2 (dose expansion cohort) of each 4 week cycle. Dose expansion cohort was added after the maximum tolerated dose (MTD) was determined from the dose limiting toxicity (DLT) evaluation.
- Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin: Study drugs were administered at following regimens in repeating 4 week cycles; Sunitinib at dose of 37.5 mg orally once daily for 2 weeks followed by 2 weeks off-treatment (Schedule 2/2), S-1 at the starting dose of 80-120 mg/day based on body surface area as a twice daily for 3 weeks followed by 1 week off-treatment, cisplatin was administered once at 60 mg/m^2 on Day 1 of each 4 week cycle.
- Sunitinib 12.5 mg CDD + S-1 + Cisplatin: Study drugs were administered at following regimens in repeating 4 week cycles; Sunitinib at dose of 12.5 mg orally once daily continuously (CDD), S-1 at the starting dose of 80-120 mg/day based on body surface area as a twice daily for 3 weeks followed by 1 week off -treatment, cisplatin was administered once at 60 mg/m^2 on Day 1 of each 4 week cycle. One participant who was assigned to the sunitinib 25 mg on CDD treatment group inadvertently took sunitinib 12.5 mg/day throughout the study, therefore this participant was analyzed separately in this group.
Period: Overall Study
Arm/Group | Sunitinib 25 mg CDD + S-1 + Cisplatin | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin | Sunitinib 12.5 mg CDD + S-1 + Cisplatin
Started | 4 | 16 | 6 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 16 | 6 | 1
Not completed — Adverse Event | 2 | 4 | 0 | 1
Not completed — Global deterioration of health status | 0 | 2 | 0 | 0
Not completed — Objective progression or relapse | 2 | 9 | 6 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib 25 mg CDD + S-1 + Cisplatin | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin | Sunitinib 12.5 mg CDD + S-1 + Cisplatin | Total
Number analyzed (Participants) | 4 | 16 | 6 | 1 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (12.8) | 56.8 (11.4) | 54.8 (16.6) | 64 (0) | 57.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 8
  Male | 2 | 13 | 4 | 0 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Cycle Dose-limiting Toxicities (DLTs)
Description: A DLT is any of a predefined set of unacceptable adverse events, regardless of cause. DLTs were assessed during the first cycle (4 weeks).
Time Frame: Cycle 1 (Baseline to Week 4)
Population: DLT Evaluation Set consisted of participants who were initially enrolled for the determination of maximam tolerated dose (MTD), and either 'experienced DLT' or 'received all of the Day 1 chemotherapy, received at least 80% of their sunitinib doses, and at least 80% of S-1 doses'.
Measure: Number; unit: participants
Groups:
- Sunitinib 25 mg 2/2 + S-1 + Cisplatin (Dose Escalation Cohort): Study drugs were administered at following regimens in repeating 4 week cycles; Sunitinib at dose of 25 mg orally once daily for 2 weeks followed by 2 weeks off-treatment (Schedule 2/2), S-1 at the starting dose of 80-120 mg/day based on body surface area as a twice daily regimen for 3 weeks followed by 1 week off-treatment, cisplatin was administered once at 60 mg/m^2 on Day 1 of each 4 week cycle.
Arm/Group | Sunitinib 25 mg CDD + S-1 + Cisplatin | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (Dose Escalation Cohort) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin
Number analyzed (Participants) | 4 | 6 | 6
participants | 2 | 1 | 3

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sunitinib, SU-012662, and Total Drug (Sunitinib + SU-012662)
Time Frame: Day 1 of Cycles 1 and 2 (pre-dose, 2, 4, 6, 8, 10, and 24 hours post-dose)
Population: Participants who received Sunitinib and had sufficient plasma concentration data for calculation of pharmacokinetic parameters
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Sunitinib 25 mg 2/2 + Cisplatin + S-1 (MTD Expansion Cohort): Subset of Sunitinib 25 mg 2/2 + Cisplatin + S-1 arm consisted of participants who were additionally enrolled after the maximum tolerated dose (MTD) of sunitinib was determined as 25 mg orally once daily for 2 weeks followed by 2 weeks off-treatment
Arm/Group | Sunitinib 25 mg 2/2 + Cisplatin + S-1 (MTD Expansion Cohort)
Number analyzed (Participants) | 7
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1: Sunitinib (Sunitinib Alone) | 14.47 (5.3414)
  Cycle 2 Day 1:Sunitinib (Sunitinib+S-1+Cisplatin) | 13.14 (3.1675)
  Cycle 1 Day 1: SU-012662 (Sunitinib Alone) | 2.487 (1.1515)
  Cycle 2 Day 1:SU-012662(Sunitinib+S-1+Cisplatin) | 2.331 (1.2943)
  Cycle1 Day 1:Total Drug (Sunitinib Alone) | 16.86 (6.3194)
  Cycle 2 Day 1:Total Drug(Sunitinib+S-1+Cisplatin) | 15.41 (3.7667)

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Sunitinib, SU-012662, and Total Drug (Sunitinib + SU-012662)
Time Frame: Day 1 of Cycles 1 and 2 (pre-dose, 2, 4, 6, 8, 10, and 24 hours post-dose)
Population: as for outcome 2
Measure: Median (Full Range); unit: hrs
Arm/Group | Sunitinib 25 mg 2/2 + Cisplatin + S-1 (MTD Expansion Cohort)
Number analyzed (Participants) | 7
hrs
  Cycle 1 Day 1: Sunitinib ( Sunitinib Alone) | 5.97 [3.83 to 8.00]
  Cycle 2 Day 1: Sunitinib (Sunitinib+S-1+Cisplatin) | 7.97 [3.97 to 9.93]
  Cycle 1 Day 1: SU-012662 ( Sunitinib Alone) | 8.00 [3.83 to 10.1]
  Cycle 2 Day 1: SU-012662 (Sunitinib+S-1+Cisplatin) | 9.25 [5.97 to 23.8]
  Cycle1 Day1:Total Drug ( Sunitinib Alone) | 5.97 [3.83 to 9.22]
  Cycle 2 Day 1:Total Drug (Sunitinib+S-1+Cisplatin) | 7.92 [3.97 to 9.25]

4. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Sunitinib, SU-012662, and Total Drug (Sunitinib + SU-012662)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Day 1 of Cycles 1 and 2 (pre-dose, 2, 4, 6, 8, 10, and 24 hours post-dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Sunitinib 25 mg 2/2 + Cisplatin + S-1 (MTD Expansion Cohort)
Number analyzed (Participants) | 7
ng*h/mL
  Cycle 1 Day 1: Sunitinib (Sunitinib Alone) | 214.6 (61.682)
  Cycle 2 Day 1: Sunitinib (Sunitinib+S-1+Cisplatin) | 211.9 (46.092)
  Cycle 1 Day 1: SU-012662 (Sunitinib Alone) | 39.77 (12.857)
  Cycle 2 Day 1: SU-012662 (Sunitinib+S-1+Cisplatin) | 44.83 (24.046)
  Cycle 1 Day 1: Total Drug (Sunitinib Alone) | 254.4 (70.913)
  Cycle 2 Day 1:Total Drug (Sunitinib+S-1+Cisplatin) | 257.0 (59.324)

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tegafur and 5-FU
Time Frame: Day 1 of Cycles 1 and 2 (pre-dose, 1, 2, 4, 6, 8, and 10 hours post-dose)
Population: Participants who received S-1 and had sufficient plasma concentration data for calculation of pharmacokinetic parameters
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All)
Number analyzed (Participants) | 5
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1: Tegafur (S-1 + Cisplatin) | 1500 (147.65)
  Cycle 2 Day 1: Tegafur (Sunitinib+S-1+Cisplatin) | 1540 (184.39)
  Cycle 1 Day 1: 5-FU (S-1 + Cisplatin) | 144.4 (33.901)
  Cycle 2 Day 1: 5-FU (Sunitinib+S-1+Cisplatin) | 105.7 (19.318)

6. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Tegafur and 5-FU
Time Frame: Day 1 of Cycles 1 and 2 (pre-dose, 1, 2, 4, 6, 8, and 10 hours post-dose)
Population: as for outcome 5
Measure: Median (Full Range); unit: hrs
Arm/Group | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All)
Number analyzed (Participants) | 5
hrs
  Cycle 1 Day 1: Tegafur (S-1 + Cisplatin) | 1.98 [0.917 to 3.98]
  Cycle 2 Day 1: Tegafur (Sunitinib+S-1+Cisplatin) | 2.00 [0.933 to 2.05]
  Cycle 1 Day 1:5-FU (S-1 + Cisplatin) | 2.00 [1.98 to 3.98]
  Cycle 2 Day 1: 5-FU (Sunitinib+S-1+Cisplatin) | 2.05 [2.00 to 4.13]

7. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Tegafur and 5-FU
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Day 1 of Cycles 1 and 2 (pre-dose, 1, 2, 4, 6, 8, and 10 hours post-dose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All)
Number analyzed (Participants) | 5
ng*h/mL
  Cycle 1 Day 1: Tegafur (S-1 + Cisplatin) | 8314 (726.38)
  Cycle 2 Day 1: Tegafur (Sunitinib+S-1+Cisplatin) | 9182 (819.65)
  Cycle 1 Day 1: 5-FU (S-1 + Cisplatin) | 582.4 (109.12)
  Cycle 2 Day 1: 5-FU (Sunitinib+S-1+Cisplatin) | 494.8 (124.14)

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Total Platinum and Free Platinum
Time Frame: Day 1 of Cycles 1 and 2 (pre-dose, 0.5, 1, 2, 8, and 22 hours after completing infusion)
Population: Participants who received cisplatin and had sufficient plasma concentration data for calculation of pharmacokinetic parameters
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All)
Number analyzed (Participants) | 5
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1: Total (S-1 + Cisplatin) | 1794 (140.11)
  Cycle 2 Day1: Total (Sunitinib+S-1+Cisplatin) | 1984 (72.319)
  Cycle 1 Day 1: Free (S-1 + Cisplatin) | 177.8 (121.47)
  Cycle 2 Day 1:Free (Sunitinib+S-1+Cisplatin) | 186.9 (139.45)

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Total Platinum and Free Platinum
Time Frame: Day 1 of Cycles 1 and 2 (pre-dose, 0.5, 1, 2, 8, and 22 hours after completing infusion)
Population: as for outcome 8
Measure: Median (Full Range); unit: hrs
Arm/Group | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All)
Number analyzed (Participants) | 5
hrs
  Cycle 1 Day 1: Total (S-1 + Cisplatin) | 2.65 [2.50 to 2.93]
  Cycle 2 Day1: Total (Sunitinib+S-1+Cisplatin) | 2.68 [2.58 to 2.90]
  Cycle 1 Day 1: Free (S-1 + Cisplatin) | 2.65 [2.50 to 2.83]
  Cycle 2 Day 1:Free (Sunitinib+S-1+Cisplatin) | 2.68 [2.58 to 2.90]

10. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Total Platinum and Free Platinum
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Day 1 of Cycles 1 and 2 (pre-dose, 0.5, 1, 2, 8, and 22 hours after completing infusion)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All)
Number analyzed (Participants) | 5
ng*h/mL
  Cycle 1 Day 1: Total (S-1 + Cisplatin) | 29020 (2070.5)
  Cycle 2 Day1: Total (Sunitinib+S-1+Cisplatin) | 33000 (2192.0)
  Cycle 1 Day 1: Free (S-1 + Cisplatin) | 967.8 (332.03)
  Cycle 2 Day 1:Free (Sunitinib+S-1+Cisplatin) | 1154 (417.55)

11. Secondary Outcome: Number of Participants With Objective Response
Description: Number of participants with objective response-based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR defined as the disappearance of all target lesions. PR defined as greater than or equal to (≥) 30 percent (%) decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. Confirmed responses are those that persist on repeat imaging at least 4 weeks after initial documentation of response.
Time Frame: Baseline up to 739 days
Population: Full Analysis Set consisted of all participants enrolled in the study who received at least 1 dose of study medication (cisplatin, S-1 or sunitinib)
Measure: Number; unit: participants
Arm/Group | Sunitinib 25 mg CDD + S-1 + Cisplatin | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin | Sunitinib 12.5 mg CDD + S-1 + Cisplatin
Number analyzed (Participants) | 4 | 16 | 6 | 1
participants | 2 | 6 | 2 | 0

12. Secondary Outcome: Number of Participants With Clinical Benefit Response (CBR)
Description: CBR is defined as a confirmed complete response (CR), confirmed partial response (PR), or stable disease (SD) for at least 24 weeks on study according to RECIST. Confirmed responses are those that persist on repeat imaging at least 4 weeks after initial documentation of response.
Time Frame: Baseline up to 739 days
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Sunitinib 25 mg CDD + S-1 + Cisplatin | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin | Sunitinib 12.5 mg CDD + S-1 + Cisplatin
Number analyzed (Participants) | 4 | 16 | 6 | 1
participants | 2 | 12 | 4 | 0

13. Secondary Outcome: Duration of Response (DR)
Description: Time from the first objective documentation of tumor response (confirmed or partial response) to first documented objective tumor progression or death due to cancer. DR calculated as (the end date for DR minus first subsequent confirmed CR or PR plus 1 day).
Time Frame: Baseline up to 739 days
Population: A subgroup of participants with an objective tumor response among Full Analysis Set consisted of all participants enrolled in the study who received at least 1 dose of study medication (cisplatin, S-1 or sunitinib)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib 25 mg CDD + S-1 + Cisplatin | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin | Sunitinib 12.5 mg CDD + S-1 + Cisplatin
Number analyzed (Participants) | 2 | 6 | 2 | 0
Months | 5.7 [5.4 to 5.9] | 10.4 [3.2 to NA] — There were too few events (objective tumor progression or death) to estimate the upper limit of confidence interval | 5.0 [4.6 to 5.3] |

14. Secondary Outcome: Progression-Free Survival (PFS)
Description: Median time from the enrollment to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first. PFS calculated as (first event date minus enrollment date plus 1 day)
Time Frame: Baseline up to 739 days
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib 25 mg CDD + S-1 + Cisplatin | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin | Sunitinib 12.5 mg CDD + S-1 + Cisplatin
Number analyzed (Participants) | 2 | 6 | 2 | 0
Months | 7.1 [6.7 to 7.5] | 12.5 [6.4 to 16.5] | 5.8 [4.4 to 7.5] |

15. Secondary Outcome: Time to Progression (TTP)
Description: Time in months from enrollment to first documentation of objective tumor progression. TTP was calculated as (first event date or last known progression-free date minus the date of enrollment plus 1 day). Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD] per RECIST).
Time Frame: Baseline up to 739 days
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib 25 mg CDD + S-1 + Cisplatin | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin | Sunitinib 12.5 mg CDD + S-1 + Cisplatin
Number analyzed (Participants) | 2 | 6 | 2 | 0
Months | 7.1 [6.7 to 7.5] | 12.5 [6.4 to 16.5] | 5.8 [4.4 to 7.5] |

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib 25 mg CDD + S-1 + Cisplatin | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin | Sunitinib 12.5 mg CDD + S-1 + Cisplatin
Serious Adverse Events (participants affected / at risk) | 2/4 | 8/16 | 2/6 | 1/1
Other Adverse Events (participants affected / at risk) | 4/4 | 16/16 | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib 25 mg CDD + S-1 + Cisplatin (N=4) | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All) (N=16) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin (N=6) | Sunitinib 12.5 mg CDD + S-1 + Cisplatin (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 2 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib 25 mg CDD + S-1 + Cisplatin (N=4) | Sunitinib 25 mg 2/2 + S-1 + Cisplatin (All) (N=16) | Sunitinib 37.5 mg 2/2 + S-1 + Cisplatin (N=6) | Sunitinib 12.5 mg CDD + S-1 + Cisplatin (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 2 | 0 | 0
Corneal disorder (Eye disorders) | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 4 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 12 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 8 | 4 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 14 | 5 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 9 | 6 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 6 | 4 | 0
Chest pain (General disorders) | 0 | 0 | 3 | 0
Extravasation (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 14 | 5 | 1
Influenza like illness (General disorders) | 0 | 3 | 2 | 0
Oedema (General disorders) | 2 | 3 | 3 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 1
Pyrexia (General disorders) | 1 | 7 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 4 | 3 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 2 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 1
Amylase increased (Investigations) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 1
Blood albumin decreased (Investigations) | 1 | 2 | 1 | 1
Blood alkaline phosphatase abnormal (Investigations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 3 | 2 | 0
Blood calcium (Investigations) | 0 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 2 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 3 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 4 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 2 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 2 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0
Glucose urine present (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 4 | 12 | 5 | 0
Lipase increased (Investigations) | 0 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 4 | 13 | 5 | 0
Platelet count decreased (Investigations) | 4 | 12 | 5 | 0
Protein total decreased (Investigations) | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 4 | 13 | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 15 | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 7 | 4 | 1
Headache (Nervous system disorders) | 0 | 2 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 5 | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 6 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 3 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 3 | 3 | 5 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.